CLINICAL TRIAL: NCT06286072
Title: The Effect of Education and Reminder Messages on the Fatigue Level of Individuals With COPD: Randomised Controlled Study
Brief Title: The Effect of Education and Reminder Messages on the Fatigue Level of Individuals With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Yasemin CEYHAN, Assistant Proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YCEYHANS
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Copd; Fatigue
Keywords: COPD; Fatigue; dyspnea; Training; Message
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fatigue; Dyspnea | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training and Message Group (Experimental): Patients in this group were given training for 3 consecutive days during their stay in the hospital.
  Day 1: general information about the disease, medication use Day 2: Physiology of fatigue, factors causing fatigue, and the relationship between COPD and fatigue.
  Day 3 Strategies to cope with fatigue (Breathing exercises, good thinking, etc.)
  Patients were messaged twice a week after they were discharged. Message sent for 8 weeks. Short, motivating and reminder messages were used. For example;
  * When I can control my shortness of breath, my fatigue level decreases significantly.
  * Excessive thinking and stress lead to more fatigue. That's why I stay away from negative thoughts.
  At the baseline and 8th weeks, the patients were interviewed again and their dyspnea and fatigue levels were measured again.
  Interventions: Other: Education and message
- Training Group (Experimental): Patients in this group were given training for 3 consecutive days during their stay in the hospital.
  Day 1: general information about the disease, medication use Day 2: Physiology of fatigue, factors causing fatigue, and the relationship between COPD and fatigue.
  Day 3 Strategies to cope with fatigue (Breathing exercises, good thinking, etc.)
  No other treatment was performed on these patients.
  At the baseline and end of 8 weeks, the patients were interviewed again and their dyspnea and fatigue levels were measured again.
  Interventions: Other: Education and message
- Routine Treatment and Care Group (Active Comparator): These patients received routine treatment and care in the clinic. No training was given. Message not sent.
  At the baseline and 8th weeks, the patients were interviewed again and their dyspnea and fatigue levels were measured again.
  Interventions: Other: Education and message

INTERVENTIONS:
Other: Education and message — COPD general education content and fatigue-specific coping strategies. Messages sent to phones

SUMMARY:
COPD is an important respiratory system disease that progresses with damage to the airways.Increased mucus secretion and thickening in the airways causes obstruction.This obstruction causes symptoms such as shortness of breath, cough, phlegm and wheezing.The most obvious problem that the emerging symptoms will cause for the patient is fatigue.Coping with fatigue is an important problem in COPD.

The main questions it aims to answer are:

1. Does the training given in COPD affect the level of fatigue?
2. Do the education given and text messages sent regarding COPD affect the level of fatigue?

In this study, patients were given informative education about COPD and ways to cope with fatigue were explained. Then, in order to increase the permanence of the training, motivational messages and short briefings were continued for 8 weeks.2 messages were sent per week. Three groups were created to reveal the effectiveness of the trainings and messages.

Group 1 was trained and messages were sent for 8 weeks. Group 2 was trained and no message was sent. Group 3 is the control group. No training has been provided other than routine maintenance.

The initial information of all groups was taken again at the end of the 8th week.

Main outcomes:

* Dyspnea severity,
* COPD general conditions and
* Fatigue level. The results obtained will be interpreted by comparing between 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD for the last 1 year
* Hospitalized for at least 3 days,
* Voluntary patients

Exclusion Criteria:

* Under 18 years old
* Over 85 years old
* Those with chronic fatigue syndrome
* Those with severe heart failure
* Those who had surgery in the last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue Level | Applied at baseline and after 8 weeks.
  Evaluated with COPD ASTHMA FATIGUE SCALE.
Dyspnea Severity | Applied at baseline and after 8 weeks.
  Evaluated with mMRC Dyspnea Scale

SECONDARY OUTCOMES:
COPD general condition | Applied at baseline and after 8 weeks.
  Evaluated with COPD ASSESSMENT QUESTIONNAIRE (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin CEYHAN, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Yasemin CEYHAN, Kırşehir, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No